CLINICAL TRIAL: NCT04203914
Title: Short Term Effect of Empagliflozin on Left Ventricular Relaxation in Non Diabetic Hypertensive Patients
Brief Title: Short Term Effect of Empagliflozin in Hypertension
Acronym: EMPHYT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, Sobngwi Eugene, Medical Advisor, Yaounde Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNO20168
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Hypertension
Keywords: Hypertension; Empagliflozin; Left ventricular diastolic function; Blood pressure
MeSH Terms: conditions — Hypertension | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Open label trial with before and after design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Empagliflozin 25mg daily add-on therapy
  Interventions: Drug: Empagliflozin Tablets

INTERVENTIONS:
Drug: Empagliflozin Tablets — Add-on 25mg once daily
  Other Names: SGLT2-i

SUMMARY:
The investigators assessed the 6-week effect of once daily 25mg SGLT2-i Empagliflozin on left ventricular diastolic function and blood pressure profile in non diabetic hypertensive patients

DETAILED DESCRIPTION:
Background: The rapid beneficial effects of Empagliflozin on cardiovascular mortality and hospitalizations rates for heart failure according to the Cardiovascular Outcome Event Trial in Type 2 Diabetes Mellitus Patients (EMPA-REG OUTCOME) trial raise some question in the mechanism of myocardial action. The investigators conducted this study in a population of non-diabetic hypertensive patients in order to look for a short-term effect on left ventricular relaxation.

Methods: The investigators carried out a single arm non- randomized clinical trial and assigned patients to receive 25mg of empagliflozin once daily in additional therapy for six weeks at the National Center for Obesity and in the cardiology department of Yaounde Central Hospital in hypertensive patients with cardiac relaxation disorder. The objectives were to evaluate the left ventricular diastolic function and nycthemeral blood pressure profile.

ELIGIBILITY:
Inclusion Criteria:

* Grade 1 hypertension
* Grade 1 or 2 relaxation abnormalities (Doppler E/A ratio <1)
* Unchanged antihypertensive treatment for at least 12 weeks

Exclusion Criteria:

* Diabetes mellitus
* eGFR < 60 mL/min/1,73 m²
* Mitral stenosis
* Atrial fibrillation
* Alanine transferase above 2N

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Left ventricular diastolic function | 6 weeks
  Doppler ultrasound measured relaxation

SECONDARY OUTCOMES:
Blood pressure | 6 weeks
  24-h ambulatory blood pressure
HbA1c | 6 weeks
  Glycated haemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Jean Claude Mbanya, MD, PhD, Study Chair — University of Yaounde 1, Cameroon; Eugene Sobngwi, MD, PhD, Principal Investigator — University of Yaounde 1, Cameroon
Locations (2):
- Cameroon (2):
  - National Obesity Centre, Yaounde Central Hospital, Yaoundé, Centre Region
  - Yaounde Central Hospital, Yaoundé, Centre Region

IPD SHARING:
Plan to Share IPD: Yes
Centrally available database available on request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 2019 for 5 years
Access Criteria: Requirements of Cameroon Ethics authorities